CLINICAL TRIAL: NCT00006481
Title: A Phase III Comparison of Biafine to Declared Institutional Preference for Radiation Induced Skin Toxicity in Patients Undergoing Radiation Therapy for Advanced Squamous Cell Carcinomas of the Head and Neck
Brief Title: Biafine Cream to Reduce Side Effects of Radiation Therapy in Patients Receiving Treatment for Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Supportive Care
Other Study IDs: RTOG-9913; CDR0000068312; NCI-P00-0173
Record Dates: First submitted 2000-11-06; First posted 2003-12-31 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2013-11

CONDITIONS: Head and Neck Cancer; Skin Reactions Secondary to Radiation Therapy
Keywords: stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; skin reactions secondary to radiation therapy
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Biafine cream
Procedure: quality-of-life assessment
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells, but may cause skin irritation and inflammation. Biafine cream may be effective in lessening side effects caused by radiation therapy.

PURPOSE: Randomized phase III trial to determine the effectiveness of Biafine cream in reducing side effects of radiation therapy in patients receiving treatment for head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of prophylactic Biafine cream vs standard best supportive care in reducing grade 2 or higher radiation-induced skin toxicity observed during radiotherapy in patients with advanced squamous cell carcinoma of the head and neck. II. Determine if prophylactic or interventional use of Biafine cream is more effective based on a reduction in maximum skin toxicity resulting from radiation treatment in this patient population. III. Compare quality of life of these patients with this treatment. IV. Assess the toxicity of Biafine cream in these patients.

OUTLINE: This is a randomized study. Patients are stratified according to lymph node status (negative vs positive), type of treatment (radiation plus chemotherapy vs radiation alone), radiation fractionation (standard vs concurrent boost), and radiation dose (50-60 Gy vs greater than 60 Gy). Patients are randomized to 1 of 3 treatment arms. Arm I: Patients receive radiotherapy once daily 5 days a week for 5-8 weeks, with or without standard skin cream application (no Biafine cream) to irradiated skin. Arm II: Patients receive radiotherapy as in arm I, with Biafine cream applied to skin 3 times daily 7 days a week at the initiation of radiotherapy and continuing for 2 weeks after the last radiation treatment. Biafine cream is applied no fewer than 4 hours before treatment and no fewer than 4 hours between applications. Arm III: Patients receive radiotherapy as in arms I and II, with Biafine cream applied as in arm II only after skin becomes symptomatic (i.e., redness, dryness, itching, or tenderness). Quality of life is assessed before treatment, weekly during treatment, and then weekly for 4 weeks after treatment completion. Patients are followed weekly for 4 weeks.

PROJECTED ACCRUAL: Approximately 500 patients will be accrued for this study within 17 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage III or IV squamous cell carcinoma of the head and neck, including: Oral cavity Oropharyngeal Hypopharyngeal Laryngeal Radiotherapy indicated as primary treatment or treatment after primary surgical resection Primary field to receive at least 50 Gy No skin rash, ulceration, or open wound in treatment field No tumor involvement of the skin

PATIENT CHARACTERISTICS: Age: Not specified Performance status: Zubrod 0-1 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: No known skin allergy or sensitivity to Biafine No inflammatory or connective tissue disorders of the skin No history of mental incompetence, including psychological disorders or drug dependency disorders, that would preclude study compliance

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: Concurrent chemotherapy allowed Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics No prior radiotherapy to treatment field Surgery: See Disease Characteristics Prior surgery allowed Other: No other concurrent investigational therapy No concurrent participation on other RTOG clinical trials No concurrent amifostine (concurrent pilocarpine allowed)

Ages: 0 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-10; Primary Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Elliott, MRT(T), MRT(R), CCRP, Study Chair — Margaret and Charles Juravinski Cancer Centre
Locations (260):
- United States (240):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Huntsville Hospital System, Huntsville, Alabama
  - Comprehensive Cancer Institute of Huntsville, Huntsville, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Alabama Oncology, LLC, Montgomery, Alabama
  - Radiation Oncology Associates of West Alabama, Tuscaloosa, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Mount Diablo Medical Center, Concord, California
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - California Cancer Center, Fresno, California
  - Saint Agnes Cancer Center, Fresno, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Sutter Health West Cancer Research Group, Greenbrae, California
  - University of California San Diego Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Huntington Cancer Center, Pasadena, California
  - Cancer Care Center, Pomona, California
  - Radiation Oncology Center - Sacramento, Sacramento, California
  - Radiation Medical Group, Inc., San Diego, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - O'Connor Hospital, San Jose, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - Saint Mary's Hospital and Medical Center, Grand Junction, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Lykes Center for Radiation Therapy, Clearwater, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - Radiation Therapy Associates - Fort Myers, Fort Myers, Florida
  - University of Florida Health Science Center, Gainesville, Florida
  - Health First Holmes Regional Medical Center, Melbourne, Florida
  - Veterans Affairs Medical Center - Miami, Miami, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Radiation Oncology Group, Orange Park, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - Sarasota Radiation and Medical Oncology Center, Sarasota, Florida
  - Tallahassee Memorial Healthcare, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical Center/John B. Amos Community Cancer Center, Columbus, Georgia
  - Regional Radiation Oncology Center at Rome, Rome, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Provena St. Joseph Hospital- Regional Cancer Care Center, Elgin, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - St. John's Medical Center, Anderson, Indiana
  - Bloomington Hospital, Bloomington, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - Clarion Health Partners Inc., Indianapolis, Indiana
  - Community Hospitals of Indianapolis - Regional Cancer Center, Indianapolis, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Louisville Radiation Oncology, Louisville, Kentucky
  - Merle M. Mahr Cancer Center, Madisonville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Romagosa Radiation Oncology Center, Lafayette, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Radiation Oncology Affiliates of Maryland, P.A., Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Regional Cancer Center, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Mary's Medical Center, Saginaw, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - North Mississippi Medical Center/Cancer Center, Tupelo, Mississippi
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Nebraska Health System, Omaha, Nebraska
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Atlantic City Medical Center, Pomona, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Associated Radiologists, P.A., Warren Township, New Jersey
  - Saint Joseph Medical Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Finger Lakes Radiation Oncology, P.C., Clifton Springs, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Beth Israel Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Vassar Brothers Hospital, Poughkeepsie, New York
  - University of Rochester Cancer Center, Rochester, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Riverhill Radiation Oncology, Yonkers, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Northeast Medical Center, Concord, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Catawba Memorial Hospital, Hickory, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Meritcare Roger Maris Cancer Center, Fargo, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - St. Anthony Hospital, Oklahoma City, Oklahoma
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - St. John Health System, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Regional Cancer Center, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Fitzgerald Mercy Hospital, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Cancer Center, East Stroudsburg, Pennsylvania
  - Penn State Geisinger Cancer Center, Hershey, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Philadelphia, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Wilkes Barre General Hospital, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Roger Williams Medical Center/BUSM, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Julie and Ben Rogers Cancer Institute, Beaumont, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall - 59th Medical Wing, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - East Texas Medical Center - Cancer Institute, Tyler, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - RMH Regional Canter Center, Harrisonburg, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Bon-Secours - St. Mary's Hospital, Richmond, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Cancer Center, Wheeling, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Foundation, La Crosse, Wisconsin
  - Southern Wisconsin Radiotherapy Center, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - St. Joseph's Hospital, Milwaukee, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - Southeastern Wisconsin Regional Cancer Center, Racine, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Canada (20):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Elliott EA, Wright JR, Swann RS, Nguyen-Tan F, Takita C, Bucci MK, Garden AS, Kim H, Hug EB, Ryu J, Greenberg M, Saxton JP, Ang K, Berk L; Radiation Therapy Oncology Group Trial 99-13. Phase III Trial of an emulsion containing trolamine for the prevention of radiation dermatitis in patients with advanced squamous cell carcinoma of the head and neck: results of Radiation Therapy Oncology Group Trial 99-13. J Clin Oncol. 2006 May 1;24(13):2092-7. doi: 10.1200/JCO.2005.04.9148. PMID 16648511